CLINICAL TRIAL: NCT04320251
Title: Tissue Growth Characterization for Cochlear Implant Users
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jack Noble, Assistant Professor, Dept. Electrical Engineering & Computer Science, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 192257
Record Dates: First submitted 2020-03-21; First posted 2020-03-24 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Cochlear Implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1 (Experimental): The single observational cohort
  Interventions: Procedure: cochlear implant revision surgery

INTERVENTIONS:
Procedure: cochlear implant revision surgery — Observation during routine cochlear implant revision surgery

SUMMARY:
It is known from post-mortem histological studies that a significant portion of individuals who undergo cochlear implantation (CI) have scar tissue form around the implanted electrode array over time. This scar tissue affects the electrical performance of the cochlear implant, affecting how the implant stimulates the auditory nerve. It is possible that if this scar tissue was detected, the implant programming could be adjusted to account for the changing tissue properties. As part of another study, a computational modeling approach for patient-customized simulation of cochlear implant stimulation is being developed. The simulation approach uses as input CT images and electrophysiological measurements from the cochlear implant device to simulate stimulation by the cochlear implant. These computational simulation models also provide a way to estimate tissue growth around the array. Tissue growth estimates are optimized in the computational model so that electrophysiological metrics simulated by the model match measurements acquired from the patient's implant. In this study, the aim is to collect data necessary to validate these model predictions.

While the existence of tissue growth around the implanted array is not typically known for most patients, a subset of cochlear implant recipients need to undergo revision surgery when a device failure or poor placement is suspected. For these individuals, the existence of tissue growth around the array in the base of the cochlea can be visualized in the operating room by the surgeon. Individuals will be recruited who are undergoing CI revision surgery at Vanderbilt University Medical Center to participate in this study. In surgery, the presence of scar tissue growth will be evaluated by visual confirmation by the surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age and above undergoing revision cochlear implant surgery.

Exclusion Criteria:

* Age < 18 years or not undergoing revision cochlear implant surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-06-15 (Estimated); Primary Completion 2027-01-09 (Estimated); Study Completion 2027-01-09 (Estimated)

PRIMARY OUTCOMES:
Tissue growth | intraoperative
  Number of individuals with observation of tissue growth around the array by cochlear implant revision surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Jack Noble, PhD, Principal Investigator — Vanderbilt University; Robert Labadie, MD,PhD, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No